CLINICAL TRIAL: NCT03727022
Title: A Phase 2, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study Evaluating the Safety and Bone Health of Multiple Injections of SM04690 Injected in the Target Knee of Moderately to Severely Symptomatic Osteoarthritis Subjects
Brief Title: Safety and Bone Health Study of SM04690 for the Treatment of Moderately to Severely Symptomatic Knee Osteoarthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biosplice Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SM04690-OA-06
Record Dates: First submitted 2018-10-30; First posted 2018-11-01 (Actual); Results first posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Knee Osteoarthritis
Keywords: SM04690; osteoarthritis; Samumed; lorecivivint; DYRK1a; CLK2
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — lorecivivint

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 0.07 mg SM04690 (Experimental): Intra-articular injections of 0.07 mg SM04690 in 2 mL vehicle
  Interventions: Drug: SM04690
- Vehicle (Placebo Comparator): Intra-articular injections of 0 mg SM04690 in 2 mL vehicle
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Healthcare professional-administered intra-articular injections; first performed on Day 1 and second at Week 24. (In the extension phase, healthcare professional-administered intra-articular injections; first performed at Week 52 and second at Week 76.)
  Other Names: vehicle
  Arms: Vehicle
Drug: SM04690 — Healthcare professional-administered intra-articular injections; first performed on Day 1 and second at Week 24. (In the extension phase, healthcare professional-administered intra-articular injections; first performed at Week 52 and second at Week 76.)
  Other Names: lorecivivint
  Arms: 0.07 mg SM04690

SUMMARY:
The primary purpose of this phase 2, placebo-controlled, double-blind, parallel group study was to provide an initial safety evaluation of two intra-articular (IA) injections of SM04690 (each at the dose of 0.07mg per 2mL injection) approximately six months apart into the target knee of moderately to severely symptomatic osteoarthritis (OA) subjects. Subjects who completed this 52-week long study were invited to enter the extension phase for an additional 52 weeks of treatment.

DETAILED DESCRIPTION:
Study SM04690-OA-06 was a multicenter, randomized, double-blind, placebo-controlled, parallel group study of a single concentration of 0.07 mg SM04690 per 2 mL injection injected into the target knee joint of moderately to severely symptomatic OA subjects at Day 1 and Week 24 (Phase A). Subjects who completed Phase A were eligible to enter the single-blind extension phase, Phase B, for an additional 52 weeks of study treatment, receiving the randomized Phase A treatment at Week 52 and again at Week 76. The study was primarily designed to assess the safety and tolerability of repeated SM04690 injections, focusing not only on AEs but also several assessments of bone density in the knee.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females between 40 and 80 years of age, inclusive, in general good health
2. Ambulatory
3. Diagnosis of femorotibial OA in the target knee by standard American College of Rheumatology (ACR) criteria at Screening Visit 1 (clinical AND radiographic criteria); OA of the knee is not to be secondary to any rheumatologic conditions (e.g., rheumatoid arthritis)
4. Pain compatible with OA of the knee(s) for at least 26 weeks prior to Screening Visit 1
5. Primary source of pain throughout the body is due to OA in the target knee
6. Daily OA knee pain diary average NRS intensity score ≥ 4 and ≤ 8 in the target knee on the 11-point (0-10) NRS scale for the 7 days immediately preceding Day 1
7. Pain NRS scores recorded for the target knee on at least 4 out of the 7 days immediately preceding Day 1
8. Daily OA knee pain diary average NRS intensity score < 4 in the non-target knee on the 11-point (0-10) NRS scale for the 7 days immediately preceding Day 1
9. Pain NRS scores recorded for the non-target knee on at least 4 out of the 7 days immediately preceding Day 1
10. WOMAC pain subscore of 20-40 (out of 50) and WOMAC physical function subscore of 68-136 (out of 170) for the target knee at baseline, regardless of if the subject is on symptomatic oral treatment (baseline questionnaire completed during the screening period prior to randomization)
11. Widespread Pain Index (WPI) score of ≤ 4 and a Symptom Severity Question 2 (SSQ2) score of ≤ 2 at Screening Visit 1
12. Willingness to use an electronic diary on a daily basis in the evening for the screening period and 104-week study duration
13. Negative drug test for amphetamine, buprenorphine, cocaine, methadone, opiates, phencyclidine (PCP), propoxyphene, barbiturates, benzodiazepine, methaqualone, and tricyclic antidepressants, except if any such drugs are clinically indicated and allowed by the protocol, at Screening Visit 1.
14. Subjects with depression or anxiety must be clinically stable for 12 weeks prior to Screening Visit 1 in the opinion of the Investigator and, if on treatment for depression or anxiety, be on 12 weeks of stable therapy
15. Full understanding of the requirements of the study and willingness to comply with all study visits and assessments
16. Subjects must have read and understood the Informed Consent Form (ICF), and must have signed and dated it prior to any study-related procedure being performed
17. Subject's Screening Visit 1 visit must occur while enrollment into the study is open
18. Subject is able to have a Screening Visit 2 qCT image acquired that does not require a re-scan as determined by the central imaging vendor

Exclusion Criteria:

1. Pregnant and breastfeeding women, and women who are not post-menopausal (defined as 12 months with no menses without an alternative medical cause) or permanently surgically sterile (includes hysterectomy, bilateral salpingectomy, and bilateral oophorectomy) and have a positive or indeterminate pregnancy result at Screening Visit 2 or Day 1
2. Women who are not post-menopausal or permanently surgically sterile, who are sexually active, and who are not willing to use birth control (as outlined in Section 5.3.1) during the study period
3. Males who are sexually active and have a partner who is capable of becoming pregnant, neither of whom have had surgery to become sterilized or who are not using birth control as outlined in Section 5.3.1
4. Body mass index (BMI) > 35
5. Partial or complete joint replacement in either knee
6. Currently requires:

   1. regular use (in the opinion of the Investigator) of ambulatory assistive devices (e.g., wheelchair, parallel bars, walker, canes, or crutches), or
   2. use of a lower extremity prosthesis, and/or a structural knee brace (i.e., a knee brace that contains hardware)
7. Radiographic disease Stage 0, 1, or 4 in the target knee at Screening Visit 1 according to the Kellgren-Lawrence grading of knee OA as assessed by independent central readers
8. Previous enrollment in a Samumed clinical trial investigating SM04690
9. Any surgery (e.g., arthroscopy) in either knee within 26 weeks prior to Screening Visit 1
10. Any bone fracture(s) within 26 weeks prior to Screening Visit 1
11. Any surgery scheduled during the study period. Non-surgical invasive procedures conducted for a diagnostic or therapeutic purpose scheduled during the study period are not prohibited.(refer to section 7.6)
12. Significant and clinically evident misalignment of either knee that would impact subject function, as determined by the Investigator
13. History of malignancy within the last 5 years; however, subjects with prior history of in situ basal or squamous cell skin cancer are eligible if completely excised. Subjects with other malignancies are eligible if they have been continuously disease free for at least 5 years prior to Screening Visit 1
14. Clinically significant abnormal screening hematology values, blood chemistry values, or urinalysis values as determined by the Investigator
15. Any condition, including laboratory findings not included in the Screening Visit 2 laboratory tests and findings in the medical history or in the pre-study assessments, that, in the opinion of the Investigator, constitutes a risk or contraindication for participation in the study or that could interfere with the study objectives, conduct, or evaluation
16. Comorbid conditions that could affect study endpoint assessments of the target knee, including, but not limited to, rheumatoid arthritis, psoriatic arthritis, systemic lupus erythematosus, gout or pseudogout, and fibromyalgia
17. Other conditions that, in the opinion of the Investigator, could affect study endpoint assessments of either knee, including, but not limited to, peripheral neuropathy (e.g., diabetic neuropathy), symptomatic hip osteoarthritis, symptomatic degenerative disc disease, and patellofemoral syndrome
18. History of mania, bipolar disorder, psychotic disorder, schizophrenia, schizoaffective disorder, major depressive disorder, or generalized anxiety disorder
19. Participation in a clinical research trial that included the receipt of an investigational product (IP) or any experimental therapeutic procedure within 26 weeks prior to Screening Visit 1, or planned participation in any such trial
20. Treatment of the target knee with intra-articular glucocorticoids (e.g., methylprednisolone) within 12 weeks prior to Screening Visit 1
21. Any intra-articular injection into the target knee with a therapeutic aim including, but not limited to, viscosupplementation (e.g., hyaluronic acid), platelet-rich plasma (PRP), and stem cell therapies within 24 weeks prior to Screening Visit 1; treatment of the target knee with intra-articular glucocorticoids greater than 12 weeks prior to Screening Visit 1 is allowed
22. Treatment with systemic (oral, intramuscular, or intravenous) glucocorticoids greater than 10 mg prednisone or the equivalent per day within 4 weeks prior to Screening Visit 1
23. Effusion of the target knee clinically requiring aspiration within 12 weeks prior to Screening Visit 1
24. Use of electrotherapy, acupuncture, and/or chiropractic treatments for knee OA within 4 weeks prior to Screening Visit 1 (refer to Appendix 1)
25. Any known active infections, including urinary tract infection, upper respiratory tract infection, sinusitis, suspicion of intra-articular infection, hepatitis B or hepatitis C infection, and/or infections that may compromise the immune system such as human immunodeficiency virus (HIV) at Day 1
26. Subjects requiring the chronic use (i.e., regular and consistent use for ≥ 12 weeks) of centrally acting analgesics (e.g., duloxetine) (refer to Appendix 1) within 12 weeks prior to Screening Visit 1
27. Subjects requiring the chronic use (i.e., regular and consistent use for ≥ 12 weeks) of anticonvulsants (not listed in Appendix 1) within 12 weeks prior to Screening Visit 1, unless used for seizure or migraine prophylaxis
28. Subjects requiring the usage of opioids >1x per week within 12 weeks prior to Screening Visit 1
29. Topical local anesthetic agents (gels, creams, or patches such as the Lidoderm patch) used for the treatment of knee OA within 7 days of Screening Visit 1
30. Any chronic condition that has not been well controlled or subjects with a chronic condition who have not maintained a stable therapeutic regimen of a prescription therapy in the opinion of the Investigator. In addition, subjects with an HbA1c >9 at Screening Visit 2 will be excluded.
31. If on NSAIDs for the treatment of OA pain, subjects who have not maintained a stable regimen in the opinion of the Investigator at Screening Visit 1
32. Any contraindications for performing DXA scans of the hips or spine including but not limited to:

    1. other radiological investigations using contrast media or radionuclides within 7 days of Screening Visit 2
    2. weight that precludes scanning at these sites
33. Subjects who have had a single or bilateral hip replacement
34. Subjects who have a current or pending disability claim, workers' compensation, or litigation(s) that may compromise response to treatment
35. Subjects who are immediate family members (spouse, parent, child, or sibling; biological or legally adopted) of personnel directly affiliated with the study at any investigative site, or are directly affiliated with the study at any investigative site
36. Subjects employed by Samumed, LLC, or any of its affiliates or development partners (that is, an employee, temporary contract worker, or designee) responsible for the conduct of the study, or who are immediate family members (spouse, parent, child, or sibling; biological or legally adopted) of said employees responsible for the conduct of the study
37. Subject has non-evaluable DXA scans of the hips or spine (i.e., pins, screws, any surgical implant, fracture, or severe degenerative changes in the region of interest), as assessed by the central imaging vendor at the time of screening

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2018-11-28 (Actual); Primary Completion 2020-09-18 (Actual); Study Completion 2021-08-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yusuf Yazici, M.D., Study Director — Biosplice Therapeutics, Inc.
Locations (12):
- United States (12):
  - Research Site, Phoenix, Arizona
  - Research Site, Canoga Park, California
  - Research Site, Carmichael, California
  - Research Site, La Mesa, California
  - Research Site, Edgewater, Florida
  - Research Site, Miami, Florida
  - Research Site, Woodstock, Georgia
  - Research Site, Kansas City, Missouri
  - Research Site, Albuquerque, New Mexico
  - Research Site, Cincinnati, Ohio
  - Research Site, Charleston, South Carolina
  - Research Site, San Angelo, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Phase A
Arm/Group | Vehicle | 0.07 mg SM04690
Started | 50 | 51
Completed | 38 | 39
Not Completed | 12 | 12
Not completed — Lost to Follow-up | 2 | 3
Not completed — Withdrawal by Subject | 10 | 9
Period: Phase B
Arm/Group | Vehicle | 0.07 mg SM04690
Started | 32 | 33
Completed | 24 | 29
Not Completed | 8 | 4
Not completed — Lost to Follow-up | 0 | 1
Not completed — Subject Non-Compliance | 1 | 0
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Site Closure | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vehicle | 0.07 mg SM04690 | Total
Number analyzed (Participants) | 50 | 51 | 101
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.5 (9.8) | 61.3 (8.4) | 60.9 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 26 | 60
  Male | 16 | 25 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 13 | 27
  Not Hispanic or Latino | 36 | 38 | 74
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 8 | 9 | 17
  White | 41 | 40 | 81
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 27.93 (4.12) | 29.30 (3.02) | 28.63 (3.65)
Kellgren-Lawrence Grade [Count of Participants; unit: Participants] — Scoring of osteoarthritis by plain radiograph. For this study, radiographs were obtained in a posterior-anterior view using a positioning device help to ensure a ~10 degree angle.
  Kellgren-Lawrence Grades 2 and 3 were included in this study:
  Grade 2 - Minimal definite osteophytes, definite narrowing of joint space Grade 3 - Moderate moderate multiple osteophytes, definite narrowing of joint space, some sclerosis and possible deformity of bone contour
  Participants
    Grade 2 | 31 | 22 | 53
    Grade 3 | 19 | 29 | 48
Medial Joint Space Width [Mean (Standard Deviation); unit: mm] — Measuring of joint space by plain radiograph. For this study, radiographs were obtained in a posterior-anterior view using a positioning device help to ensure a ~10 degree angle. Measurement of joint space was performed by blinded central reader using a proprietary landmark algorithm.
  mm | 3.193 (1.348) | 3.119 (1.216) | 3.156 (1.277)

OUTCOME MEASURES:

1. Primary Outcome: Change in Total BMD From Baseline in the Treated Knee Compared to Placebo by qCT
Description: Evaluate change in total bone mineral density (BMD) from baseline in the treated knee compared to placebo by quantitative computed tomography (qCT)
Time Frame: Baseline and Week 52
Population: Full Analysis Set includes all subjects who received at least one study injection in Phase A. Subjects' observed data were analyzed as randomized for the FAS without imputation.
Measure: Mean (Standard Deviation); unit: mg/cm^3
Arm/Group | Vehicle | 0.07 mg SM04690
Number analyzed (Participants) | 34 | 37
mg/cm^3 | -0.47 (8.21) | -3.32 (10.00)
Statistical Analysis 1: Comparison: Vehicle vs 0.07 mg SM04690; Test type: Superiority; Mean Difference (Final Values) = -2.81, 95% CI 2-sided [-7.19 to 1.58]

2. Secondary Outcome: Change in Total BMD From Baseline in the Treated Knee Compared to Placebo by qCT
Description: Evaluate change in total BMD from baseline in the treated knee compared to placebo by qCT
Time Frame: Baseline and Weeks 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/cm^3
Arm/Group | Vehicle | 0.07 mg SM04690
Number analyzed (Participants) | 43 | 45
mg/cm^3 | -0.38 (7.89) | -0.34 (7.28)
Statistical Analysis 1: Comparison: Vehicle vs 0.07 mg SM04690; Test type: Superiority; Mean Difference (Final Values) = -0.00, 95% CI 2-sided [-3.24 to 3.24]

3. Secondary Outcome: Change in Total BMD From Baseline in the Treated Knee Compared to Placebo by qCT
Description: Evaluate change in total BMD from baseline in the treated knee compared to placebo by qCT
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/cm^3
Arm/Group | Vehicle | 0.07 mg SM04690
Number analyzed (Participants) | 40 | 39
mg/cm^3 | 1.34 (7.77) | -0.76 (8.81)
Statistical Analysis 1: Comparison: Vehicle vs 0.07 mg SM04690; Test type: Superiority; Mean Difference (Final Values) = -2.09, 95% CI 2-sided [-5.84 to 1.65]

4. Secondary Outcome: Change in Total BMD From Baseline in the Treated Knee Compared to Placebo by qCT
Description: Evaluate change in total BMD from baseline in the treated knee compared to placebo by qCT
Time Frame: Baseline and Week 36
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/cm^3
Arm/Group | Vehicle | 0.07 mg SM04690
Number analyzed (Participants) | 36 | 33
mg/cm^3 | -1.82 (8.47) | -2.06 (7.18)
Statistical Analysis 1: Comparison: Vehicle vs 0.07 mg SM04690; Test type: Superiority; Median Difference (Final Values) = -0.25, 95% CI 2-sided [-4.05 to 3.54]

5. Secondary Outcome: Change in Total BMD From Baseline in the Treated Knee Compared to Placebo by qCT
Description: as for outcome 1
Time Frame: Baseline and Week 64
Population: Full Analysis Set (FASB) includes all subjects who received at least one study injection in Phase B. Subjects' observed data were analyzed as randomized for the FASB without imputation.
Measure: Mean (Standard Deviation); unit: mg/cm^3
Arm/Group | Vehicle | 0.07 mg SM04690
Number analyzed (Participants) | 25 | 30
mg/cm^3 | -4.56 (9.84) | -3.76 (9.94)
Statistical Analysis 1: Comparison: Vehicle vs 0.07 mg SM04690; Test type: Superiority; Mean Difference (Final Values) = 0.80, 95% CI 2-sided [-4.64 to 6.23]

6. Secondary Outcome: Change in Total BMD From Baseline in the Treated Knee Compared to Placebo by qCT
Description: Evaluate change in total BMD from baseline in the treated knee compared to placebo by qCT
Time Frame: Baseline and Week 76
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mg/cm^3
Arm/Group | Vehicle | 0.07 mg SM04690
Number analyzed (Participants) | 25 | 30
mg/cm^3 | -2.13 (8.94) | -5.61 (10.67)
Statistical Analysis 1: Comparison: Vehicle vs 0.07 mg SM04690; Test type: Superiority; Mean Difference (Final Values) = -3.2, 95% CI 2-sided [-8.64 to 2.23]

7. Secondary Outcome: Change in Total BMD From Baseline in the Treated Knee Compared to Placebo by qCT
Description: Evaluate change in total BMD from baseline in the treated knee compared to placebo by qCT
Time Frame: Baseline and Week 88
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mg/cm^3
Arm/Group | Vehicle | 0.07 mg SM04690
Number analyzed (Participants) | 23 | 28
mg/cm^3 | -2.59 (10.52) | -5.14 (11.59)
Statistical Analysis 1: Comparison: Vehicle vs 0.07 mg SM04690; Test type: Superiority; Mean Difference (Final Values) = -2.36, 95% CI 2-sided [-8.75 to 4.03]

8. Secondary Outcome: Change in Total BMD From Baseline in the Treated Knee Compared to Placebo by qCT
Description: Evaluate change in total BMD from baseline in the treated knee compared to placebo by qCT
Time Frame: Baseline and Week 104
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mg/cm^3
Arm/Group | Vehicle | 0.07 mg SM04690
Number analyzed (Participants) | 24 | 29
mg/cm^3 | -2.95 (13.21) | -7.08 (12.34)
Statistical Analysis 1: Comparison: Vehicle vs 0.07 mg SM04690; Test type: Superiority; Median Difference (Final Values) = -4.05, 95% CI 2-sided [-11.21 to 3.11]

ADVERSE EVENTS:
Time Frame: Baseline to End of Study Visit at Week 104 (2 years)
Arm/Group | 0.07 mg SM04690 | Vehicle
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/50
Serious Adverse Events (participants affected / at risk) | 2/51 | 2/50
Other Adverse Events (participants affected / at risk) | 11/51 | 14/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.07 mg SM04690 (N=51) | Vehicle (N=50)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hormone receptor positive breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Intracranial aneurysm (Nervous system disorders) | 1 (1) | 0 (0)
Aortic valve incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Nodal rhythm (Cardiac disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Procedural pneumothorax (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.07 mg SM04690 (N=51) | Vehicle (N=50)
Blood pressure increased (Investigations) | 4 (4) | 1 (2)
Sinusitis (Infections and infestations) | 3 (4) | 1 (1)
COVID-19 (Infections and infestations) | 2 (2) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (5)
Nasopharyngitis (Infections and infestations) | 1 (1) | 2 (2)
Cerumen impaction (Ear and labyrinth disorders) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There is an agreement between the Principal Investigator and the Sponsor (or its agents) that restricts the PI's rights to discuss or publish trial results after the trial is completed.

DOCUMENTS (2):
  • Study Protocol (2020-08-21): https://cdn.clinicaltrials.gov/large-docs/22/NCT03727022/Prot_001.pdf
  • Statistical Analysis Plan (2021-09-22): https://cdn.clinicaltrials.gov/large-docs/22/NCT03727022/SAP_002.pdf